CLINICAL TRIAL: NCT01816828
Title: A Small Group Intervention to Reduce HIV Sexual Transmission Risk Behaviour Among HIV Positive Men Who Have Sex With Men: Gay Poz Sex (GPS)
Brief Title: Intervention Research to Reduce HIV Sexual Transmission Among HIV Positive Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: University of Windsor (Other); Simon Fraser University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Trevor Hart, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DCO150GP
Record Dates: First submitted 2013-03-19; First posted 2013-03-22 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: HIV
Keywords: HIV, MSM, unprotected anal intercourse, sexual health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate (Experimental): In the immediate arm, participants will begin the 8 session group motivational interviewing intervention, Gay Poz Sex, within 2 weeks of randomization.
  Interventions: Behavioral: Gay Poz Sex
- Wait List/Standard of Care (Active Comparator): Participants in the wait list/standard of care group will be given active referrals to existing community resources available to HIV+ MSM. For ethical reasons, participants randomized to the control group will have the option to attend the Gay Poz Sex program after a 6-month wait period.
  Interventions: Other: Wait List/Standard of Care

INTERVENTIONS:
Behavioral: Gay Poz Sex — Gay Poz Sex is a community-driven, peer-facilitated program for HIV+ gay and bisexual men. This eight week program is offered to small groups of 5-8 men and provides information about sexual health, the legal context of HIV non-disclosure and uses motivational interviewing to support each individual in setting and achieving a personal goal.
  Arms: Immediate
Other: Wait List/Standard of Care — Participants are given referrals to existing resources in the community. Referrals and uptake will be tracked.
  Arms: Wait List/Standard of Care

SUMMARY:
Gay Poz Sex (GPS) is a peer-facilitated holistic sexual health program for gay and bisexual HIV-positive men. Groups of five to eight men attend eight weekly sessions which cover basic sexual health information, review the current legal context surrounding HIV non-disclosure and use motivational interviewing (MI) to support participants in setting and achieving personal goals.

In this randomized control trial phase of the research, the investigators are assessing the efficacy of the group counseling intervention, GPS. Participants are randomized to receive GPS immediately or to a wait list/standard of care condition. Participants are followed for a 6 month period and are asked to complete baseline quantitative assessments, as well as two qualitative interviews.

DETAILED DESCRIPTION:
The randomized control trial (RCT) component will test the efficacy of GPS, an HIV prevention intervention for HIV+ men who have sex with men (MSM). The present study is intended to be a rigorous evaluation, with the ultimate aim of testing the scale-up of the GPS program using a Phase IV effectiveness trial, per standard procedures for evaluating health interventions. The study hypothesis is that the study intervention will result in reduced prevalence of unprotected anal intercourse (UAI) acts among HIV+ MSM at 6-month follow-up with partners who are negative or of unknown HIV status. The secondary hypotheses are that the intervention will result in (1) reduced prevalence of UAI at 6-months follow-up with partners who are HIV+, and (2) a reduction in the number of sexual partners.

This is a 2-site, 2-arm, randomized controlled trial that will randomize 180 participants to either a 8 session group motivational interviewing intervention (GPS) starting within 2 weeks after randomization, or to a wait-list control group. For ethical reasons, participants randomized to the control group will have the option to attend a GPS session after a 6-month wait period. Participants will complete 8 sessions of a small-group sexual health intervention to reduce sexual risk behaviour. Assessments will be conducted prior to the 8-session group, at the completion of the sessions and at 3-month and 6-month follow up post-intervention. The wait-list control group will complete 3- and 6-month follow-up assessments during their waiting period as well as after completing their GPS session. The 6 month follow-up assessment during their waiting period will be considered to be the baseline measure for their GPS session. Participants in both groups will complete interviews at the end of the 8 sessions and at the 6-month follow up.

GPS takes the form of a small counseling group, since this is one of the most common intervention forms for similar populations. Participants will be organized into 15 groups per arm of approximately 6 participants, each of which will be led by 2 facilitators who are HIV+ MSM. This study builds upon a one-armed open-label Canadian Institutes for Health Research (CIHR)-funded grant that demonstrated that GPS is feasible to administer and appears to result in significant risk reduction. The study also showed that GPS results in promising reductions in UAI, thus forming a solid foundation for moving toward an RCT. In preliminary GPS data (n=25), we found a reduction in UAI from 88% at baseline to 60% at 3-month follow-up. More importantly for HIV prevention, we found a reduction in UAI with partners of HIV-negative or unknown HIV status from 56% at baseline to 36% at 6 month follow-up. Participants reported high satisfaction with the GPS program and our initial study site has found GPS to be highly feasible in their community organization.

The proposed study will provide data on the efficacy of a motivational interviewing behavioural intervention for HIV+ MSM. Although research among primarily American samples documents moderate effect sizes for HIV prevention interventions among MSM, none have found a significant effect of an HIV prevention intervention for HIV+ MSM in Canada, nor have any studies examined the effect of a small-group based intervention using HIV+ MSM peers who are trained to administer motivational interviewing for HIV+ MSM. Armed with the data from the present study demonstrating the efficacy of the intervention, we will design and implement the next stage of the research program, which will be a Phase IV study to examine the effectiveness of the intervention in Toronto, Vancouver, and at least 2 other sites serving HIV+ MSM in Canada.

The intervention should result in a decreased likelihood of having risky sex versus being on a waitlist. Previous data from formative research with this same intervention indicates promising findings that indicate a decreased prevalence of risky sex amongst GPS participants.

ELIGIBILITY:
Inclusion Criteria:

* Are an HIV-positive man who reports unprotected anal intercourse in the past two months
* Speak and understand English
* Anticipate that you will be able to attend all workshops
* Are willing to participate in program monitoring and evaluation

Exclusion Criteria:

* Currently participating in counseling using motivational interviewing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2013-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
number of UAI acts with HIV-negative or status unknown partners | 2 months
  The main outcome measure for the GPS study is number of UAI acts with HIV-negative or status unknown partners reported by HIV+ MSM participants within the past 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Trevor A Hart, PhD, Principal Investigator — Toronto Metropolitan University; Barry D Adam, PhD, Principal Investigator — Windsor University
Locations (2):
- Canada (2):
  - Positive Living Society of British Columbia, Vancouver, British Columbia
  - Ryerson University, Toronto, Ontario